CLINICAL TRIAL: NCT04393831
Title: A Prospective Trial on Nerve Sparing Techniques Performed in Radical Prostatectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated to facilitate accrual under NCT05155501
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1512016820
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer; Quality of Life
Keywords: prostate cancer; radical prostatectomy; robot-assisted radical prostatectomy; prostatectomy; nerve sparing; Retzius; quality of life; urinary incontinence; sexual function
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing Retzius sparing robot-assisted radical prostatectomy versus conventional robot-assisted radical prostatectomy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retzius sparing (Active Comparator): Using the Retzius technique, the surgeon will remove the prostate in a way that preserves a portion of the nerves and tissue structures that are typically removed during the conventional technique.
  Interventions: Procedure: Retzius sparing
- Conventional (non-Retzius) nerve sparing (No Intervention): A non-Retzius nerve sparing technique will be performed, according to surgeon's preference--nerve sparing during radical prostatectomy is performed with significant variation and there is an absence of universally agreed upon steps or techniques.

INTERVENTIONS:
Procedure: Retzius sparing — Retzius nerve sparing is a specific approach that avoids disrupting the structures involved in urinary and sexual function.
  Arms: Retzius sparing

SUMMARY:
The investigators propose a prospective study to assess recovery of urinary and sexual function by nerve sparing techniques after radical prostatectomy.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to Retzius nerve sparing versus non-Retzius nerve sparing to compare cancer outcomes and urinary/sexual outcomes following radical prostatectomy. Using the Retzius technique, the surgeon will remove the prostate in a way that preserves a portion of the nerves and tissue structures that are typically removed during the conventional technique.

The investigators will assess recovery of urinary and sexual function of patients through questionnaires at 1 week, 1 month, 6 months, 12 months, and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* clinically localized prostate cancer
* able to read and speak English or Spanish
* no previous history of head injury, dementia or psychiatric illness
* no other concurrent cancer
* estimated life expectancy of 10 years or more
* biopsy proven prostate cancer

Exclusion Criteria:

* evidence of metastases
* Prostate specific antigen (PSA) greater than 30 ng/mL
* previous major pelvic surgery
* diagnosis of another malignancy within the past 5 years, with the exception of non-melanoma skin cancer

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Related Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to 24 months following surgery
  The investigators will obtain patient-reported complications and adverse events captured from patient's medical record.
Change in Patient-reported Health-Related Quality of Life (HRQOL) Scores as Assessed by Expanded Prostate Cancer Index Composite for Clinical Practice (EPIC-CP) | Baseline, 1 month, 6 months, 12 months, and 24 months post-surgery
  Patients will fill out the EPIC-CP questionnaire. The EPIC-CP is a 10-item questionnaire assessing five health-related quality of life domains: urinary function, urinary irritation, bowel function, sexual function, and hormonal issues. All questions are about patients' health and symptoms in the last four weeks.
  Each domain is scored out of 12 points, with higher scores indicating more complications.
  In total, the EPIC-CP score is the final sum of the 5 domains. The EPIC-CP is scored out of 60 points, with higher scores indicating more issues related to overall prostate cancer quality of life.
Change from Baseline in Prostate Specific Antigen (PSA) value on Laboratory Reports up to 24 Months Following Surgery | Baseline and up to 24 months post-surgery
  The investigators will obtain patient's PSA values from their medical record, at baseline and up to 24 months post-surgery. Patient PSA levels are obtained from standard of care blood tests, and PSA values are measured in ng/mL.

SECONDARY OUTCOMES:
Change in Baseline in Patient-Reported Penile Shortening as Assessed on Questionnaire | Baseline, 1 month, 6 months, 12 months, and 24 months post-surgery
  Patients will fill out a validated, 5-item questionnaire assessing penile shortening, self-esteem, and presence of erections.
  Question 1 assesses patients' perceived penile length post-surgery, compared to penile length at 30 years of age. It consists of two possible responses: Yes or No.
  Questions 2 and 3 assesses patients' ability to obtain and quality of spontaneous morning erections and sexual activity-related erections. It consists of five possible responses: ranging from "No erections" to "Erections always sufficient".
  Question 4 is a visual digital scale assessing patients' present quality of life. It is scored on a scale of 1-7, with higher scores indicating high quality of life.
  Question 5 is a visual digital scale assessing patients' present self-esteem. It is scored on a scale of 1-7, with higher scores indicating high self-esteem.
Change in Baseline in Patient-Reported Penile Deformity as Assessed on Questionnaire | Baseline, 6 months, 12 months, and 24 months post-surgery
  Patients will fill out a validated, 3-item questionnaire assessing presence of Peyronie's disease.
  Question 1 assesses penile hardening in the flaccid state. Question 2 assesses penile curvature in the erect state. Question 3 assesses pain associated with erection. Each question consists of two possible responses: Yes or No.
Change in Patient-reported Treatment Regret Scores as Assessed by Questionnaire | 12 months, 24 months post-surgery
  Patients will fill out a validated, 5-item questionnaire assessing feelings toward treatment regret.
  Each item is scored on a 5 point scale ranging from "Strongly Agree" to "Strongly Disagree". Responses are converted to a score ranging from 0-100, with higher scores indicating more regret.

CONTACTS AND LOCATIONS:
Overall Officials: Jim C Hu, MD MPH, Principal Investigator — Weill Cornell Medicine, NewYork-Presbyterian
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.